CLINICAL TRIAL: NCT06869564
Title: Evaluation of the Discriminative Abilities of Biomarkers for the Diagnosis of Acute Mesenteric Ischemia Compared With Another Similar Clinical Presentation: a Pilot Study
Acronym: SOS-ISMES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RCAPHM24_0416; 2024-A02484-43 (Other: IDRCB)
Record Dates: First submitted 2025-02-26; First posted 2025-03-11 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-07

CONDITIONS: Acute Mesenteric Ischemia
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Soluble adenosine deaminase assay for the diagnosis of IMA (Experimental): Assess the overall discriminatory performance of soluble adenosine deaminase in the diagnosis of IMA, compared with the reference method (injected abdominopelvic CT scan). The area under the ROC curve will be estimated, together with its 95% confidence interval.
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — At the time of blood sampling for biological tests, 2 additional tubes of blood will be taken.

SUMMARY:
Acute mesenteric ischemia (AMI) is associated with high mortality (50-80%). The prognosis depends on the time it takes to diagnose the condition, and the possibility of revascularization in eligible patients. Delayed diagnosis is due in particular to the aspecific clinical presentation and the absence of biomarkers to guide early diagnosis, lactates often being elevated at an already irreversible stage. Adenosine deaminase is produced in the presence of ischemia (known from myocardial ischemia), and is present on the surface of intestinal villi. The investigator's hypothesis is that, in the event of digestive ischemia resulting in abnormalities of mesenteric permeability, adenosine deaminase will enter the bloodstream and increase its soluble plasma activity, along with an increase in lymphocyte-bound adenosine deaminase.

The main objective is to evaluate the discriminatory capacities of soluble adenosine deaminase, collected via blood sampling, for the diagnosis of IMA in comparison with the reference method (injected abdominopelvic CT scan), performed for abdominal pain suggestive of IMA.

The study will be based on a prospective monocentric cohort. Currently, there is no specific biological marker for IMA, and the gold standard for diagnosis is the injected abdominopelvic CT scan, performed for hyperintense abdominal pain.

Two groups will be identified on the basis of the gold-standard abdominopelvic scan:

* the "IMA patients" group: patients with hyperintense abdominal pain, and IMA confirmed by CT scan
* the "non-IMA patients" group: patients with hyperintense abdominal pain, but with a diagnosis other than IMA on the CT scan.

  130 subjects will be included in this study Inclusion period: 18 months Follow-up period: 1 month Analysis period: 5 months Total duration: 24 months

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older
* with an indication (hyperintense abdominal pain with no obvious diagnosis other than acute mesenteric ischemia) for an injected abdominopelvic scan for hyperintense abdominal pain suspected of acute mesenteric ischemia
* Including pregnant or breast-feeding women, as this is a risk factor for AMI in young subjects
* Affiliated with the French social security system
* Able to express non-opposition in writing

Exclusion Criteria:

* Presenting acute myocardial ischemia, to avoid biasing the levels of the biomarkers studied (increased in this clinical situation)
* Patient in a period of exclusion from another research protocol at the time the non-opposition is signed,
* Person protected by articles L1121-6 and L1121-8 of the French Public Health Code (deprived of liberty by court order, socially vulnerable, adult incapable or unable to express non-opposition).
* Persons who are unable to read and understand the French language sufficiently to give their consent to participate in research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-06-29 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Identify soluble adenosine deaminase as a marker for the diagnosis of IMA | through study completion, an average of 2 years
  In comparison with the reference method (injected abdominopelvic CT scan), identification of soluble adenosine deaminase as a marker for the diagnosis of IMA.

SECONDARY OUTCOMES:
Rate of lymphocyte adenosine deaminase and ischemia-modified albumin | through study completion, an average of 2 years
  To evaluate the discriminative abilities of lymphocyte adenosine deaminase and ischemia-modified albumin for the diagnosis of IMA in comparison with the reference method (injected abdominopelvic CT).
threshold estimation for each biomarker | through study completion, an average of 2 years
  Determine the best threshold for each biomarker to diagnose patients with AMI.
Estimate the discriminant performance associated with the threshold selected for each biomarker. | through study completion, an average of 2 years
  Estimate the discriminant performance associated with the threshold selected for each biomarker: sensitivity, specificity, positive predictive value, negative predictive value, positive likelihood ratio, negative likelihood ratio, and their 95% confidence intervals
Description of a biological signature for IMA, including the different biomarkers measured specifically and those usually measured. | through study completion, an average of 2 years
  Biological signature of IMA including lymphocyte adenosine deaminase, soluble adenosine deaminase, ischemia-modified albumin, lactates, amylase, CPK, LDH, ASAT, CRP and D dimers
Measurement of the extent of digestive resection leaving in place the equivalent of a short small bowel (<1.5m after the duodenum) | through study completion, an average of 2 years
  Compare the rates of each of the biomarkers tested as a function of AMI severity among patients with a CT-confirmed diagnosis of AMI.
30-day prognosis | through study completion, an average of 2 years
  To compare the levels of each of the biomarkers tested in relation to the 30-day prognosis of AMI among patients with a CT-confirmed diagnosis of AMI.

CONTACTS AND LOCATIONS:
Locations (1):
- Timone hospital, Marseille, France